CLINICAL TRIAL: NCT03202979
Title: Efficacy and Safety of Low Doses of Trazodone in Patients Affected by Painful Diabetic Neuropathy: Randomized, Controlled, Pilot Study.
Brief Title: Trazodone in Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Chiltern International Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 039(B)PO16143; 2016-002772-27 (EudraCT Number)
Record Dates: First submitted 2017-06-23; First posted 2017-06-29 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Painful Diabetic Neuropathy
Keywords: Trazodone; Placebo; Gabapentin; Neuropathic pain
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia | interventions — Trazodone

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo controlled, double-dummy, dose finding, multicentre, international, prospective, pilot study.
Who Masked: Participant, Investigator
Masking Description: The present study will be performed in double blind conditions. During the study, neither the Investigator nor the patient will be aware of the treatment assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Trazodone 20 mg
  Interventions: Drug: Trazodone 20 mg
- Group 2 (Experimental): Trazodone 10 mg
  Interventions: Drug: Trazodone 10 mg
- Group 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trazodone 20 mg — Oral administration of trazodone 20 mg (corresponding to 10 drops of trazodone hydrochloride 6% oral solution), three times a day, for 8 weeks. Trazodone total daily dose: 60 mg.
  After the 8-week treatment period, patients will receive trazodone 10 mg (corresponding to 5 drops of trazodone hydrochloride 6% oral solution) three times a day for 1-week tapering period in double blind conditions.
  Other Names: Trittico®
  Arms: Group 1
Drug: Trazodone 10 mg — Oral administration of trazodone 10 mg (corresponding to 5 drops of trazodone hydrochloride 6% oral solution), three times a day, for 8 weeks. Trazodone total daily dose: 30 mg.
  In order to maintain the study double-blind conditions,patients randomized in this group will be co-administered with placebo oral solution (5 drops).
  After the 8-week treatment period, patients will receive placebo oral solution three times a day for 1-week tapering period in double blind conditions.
  Other Names: Trittico®
  Arms: Group 2
Drug: Placebo — Oral administration of placebo oral solution (10 drops) three times a day, for 8-week treatment.
  After the 8-week treatment period, patients will receive placebo oral solution three times a day for 1-week tapering period in double blind conditions.
  Arms: Group 3

SUMMARY:
The aim of the study is to collect preliminary information on the effect of low doses of trazodone on pain intensity in patients with painful diabetic neuropathy and to evaluate the neuropathic pain symptoms, anxiety, sleep, quality of life, safety and tolerability.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled, double-dummy, dose finding, parallel group, multicentre, international, prospective, pilot study.

The present study is planned to assess the efficacy and the safety of an 8-week treatment period with low doses of trazodone (30 mg daily or 60 mg total daily, respectively) administered to patients affected by painful diabetic neuropathy.

Gabapentin will be administered together with the investigational drug in open label conditions in order to assure an effective pharmacological treatment to all patients. A slow titration of gabapentin will be applied in this trial in order to control possible side effects when co-administered with trazodone.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patient of any ethnic origin between 18 and 75 years of age (limits included).
2. Patient with painful diabetic symmetric polyneuropathy manifesting with distally distributed neuropathic pain.
3. Stable glycaemic control with a value of HbA1c ≤ 10% at Screening Visit.
4. Pain persisting for at least 3 months.
5. Neuropathic pain confirmed by DN4 score ≥ 4 at Screening Visit.
6. BPI-SF 24-hour average pain score (item 5) ≥ 4 at Screening Visit and Baseline Visit.
7. Patient who is currently not receiving treatment for diabetic neuropathic pain or patient who is receiving treatment, with drug/s other than gabapentin, and have completed the required washout.
8. Women of childbearing potential must have a negative pregnancy test at Screening Visit and have to agree not to start a pregnancy from the signature of the informed consent up to thirty days after the last administration of the investigational product, using an appropriate birth control method, such as combined estrogen and progestogen containing hormonal contraception (e.g. oral, intravaginal, transdermal), progestogen-only hormonal contraception (e.g. oral, injectable, implantable), intrauterine device (IUD) or intrauterine hormone- releasing system (IUS) in combination with male condom, bilateral tubal occlusion, vasectomised partner, sexual abstinence.
9. Legally capable to give their consent to participate in the study and available to sign and date the written informed consent.

Exclusion Criteria:

1. Known hypersensitivity to trazodone or gabapentin or their excipients.
2. Other forms of neuropathic pain or non-neuropathic pain (included but not limited to peripheral arterial disease, radiculopathy, mononeuropathy, proximal motor neuropathy, post-operative pain, etc).
3. Concomitant treatment with other medications for pain management.
4. Concomitant treatment with potent CYP3A4 inhibitors (e.g. ketoconazole, ritonavir, indinavir) or drugs known to prolong QT interval.
5. Use of trazodone or gabapentin in the previous 3 months.
6. Clinically significant abnormalities on physical examination, vital signs, ECG, laboratory tests at Screening Visit that in the opinion of Investigator would compromise patient's participation in the study.
7. Active foot ulcer or previous major limb amputation.
8. Myocardial infarction or angioplasty or by-pass graft procedures within the past 6 months.
9. Patient with increased risk of Torsade de Pointes (e.g. family history of long QT syndrome) or QTcF value higher than 450 msec (male) and QTcF value higher than 470 msec (female) at Screening Visit.
10. Transient ischemic attack or cerebral vascular accident within the past 6 months.
11. GFR value < 60 ml/min calculated with MDRD formula.
12. Significant liver disease, defined as known active hepatitis or elevated liver enzymes over 3 fold the upper normal limit of laboratory normal ranges.
13. Patient with latent or known hereditary problems of galactose intolerance or the Lapp lactase deficiency or glucose-galactose malabsorption.
14. Positive urine drug screen for CNS active drugs (cocaine, opioids, amphetamines and cannabinoids) a Screening Visit.
15. Positive present history of glaucoma.
16. Hyperthyroidism, even if pharmacologically corrected.
17. Significant mental disorders.
18. History of seizure events other than a single childhood febrile seizure.
19. History of alcohol or psychoactive substance abuse or addiction.
20. Patient suffering from adrenal hypofunction (e.g. Addison's disease).
21. Women during pregnancy or lactation period.
22. Inability to comply with the protocol requirements, instructions or study-related restrictions (e.g. uncooperative attitude, inability to return for study-visits, improbability of completing the clinical study, etc).
23. Subject involved in the conduct of the study (e.g. Investigator or his/her deputy, first grade relatives, pharmacist, assistant or other personnel, etc).
24. Participation to an interventional clinical trial within 3 months prior to Screening Visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
Change of item 5 score in Brief Pain Inventory Short Form (BPI-SF) scale | Baseline - Day 56
  Change from baseline of item 5 score in BPI-SF numering scale after 56 days.

SECONDARY OUTCOMES:
Change of item 5 score in Brief Pain Inventory Short Form (BPI-SF) scale | Baseline - Days 7, 14, 21, 28, 35, 42, 49, 63
  Change from baseline of item 5 score in BPI-SF numering scale after 7, 14, 21, 28, 35, 42, 49 and 63 days.
Change of item 3 score in Brief Pain Inventory Short Form (BPI-SF) scale | Baseline - Days 7, 14, 21, 28, 35, 42, 49, 56 and 63.
  Change from baseline of item 3 score in BPI-SF numering scale after 7, 14, 21, 28, 35, 42, 49, 56 and 63 days.
Change of item 4 score in Brief Pain Inventory Short Form (BPI-SF) scale | Baseline - Days 7, 14, 21, 28, 35, 42, 49, 56 and 63.
  Change from baseline of item 4 score in BPI-SF numering scale after 7, 14, 21, 28, 35, 42, 49, 56 and 63 days.
Change of item 5 score in Brief Pain Inventory Short Form (BPI-SF) scale | Baseline - Days 7, 14, 21, 28, 35, 42, 49, 56 and 63.
  Change from baseline of item 5 score in BPI-SF numering scale after 7, 14, 21, 28, 35, 42, 49, 56 and 63 days.
Change of item 6 score in Brief Pain Inventory Short Form (BPI-SF) scale | Baseline - Days 7, 14, 21, 28, 35, 42, 49, 56 and 63.
  Change from baseline of item 6 score in BPI-SF numering scale after 7, 14, 21, 28, 35, 42, 49, 56 and 63 days.
Change of item 8 score in Brief Pain Inventory Short Form (BPI-SF) scale | Baseline - Days 7, 14, 21, 28, 35, 42, 49, 56 and 63.
  Change from baseline of item 8 score in BPI-SF numering scale after 7, 14, 21, 28, 35, 42, 49, 56 and 63 days.
Change of item 9 score in Brief Pain Inventory Short Form (BPI-SF) scale | Baseline - Days 7, 14, 21, 28, 35, 42, 49, 56 and 63.
  Change from baseline of item 9 score in BPI-SF numering scale after 7, 14, 21, 28, 35, 42, 49, 56 and 63 days.
Change in Neuropathic Pain Symptom Inventory (NPSI) scale | Baseline - Days 7, 14, 21, 28, 35, 42, 49, 56 and 63.
  Change from baseline of total score in NPSI scale after 7, 14, 21, 28, 35, 42, 49, 56 and 63 days.
Change in 36-item Short-Form Health Survey (SF-36) | Baseline - Day 56
  Change from baseline of SF-36 after 56 days.
Change in Hamilton Anxiety Rating Scale (HAM-A) | Baseline - Days 7, 14, 21, 28, 35, 42, 49, 56 and 63.
  Change from baseline of total score in HAM-A scale after 7, 14, 21, 28, 35, 42, 49, 56 and 63 days.
Patient Global Impression of Change (PGIC) | Days 7, 14, 21, 28, 35, 42, 49, 56 and 63.
  Assessment by patient of the overall efficacy and tolerability by PGIC after 7, 14, 21, 28, 35, 42, 49, 56 and 63 days
Change in Leeds Sleep Evaluation Questionnaire (LSEQ) | Baseline - Days 7, 14, 21, 28, 35, 42, 49, 56 and 63.
  Change from baseline in LSEQ after 7, 14, 21, 28, 35, 42, 49, 56 and 63 days.
Frequency of treatment-related adverse events | 9 weeks
  Monitoring of the frequency of adverse events, physical examination, vital signs, ECG, laboratory analyses

CONTACTS AND LOCATIONS:
Locations (20):
- Czechia (7):
  - NEUROHK s.r.o., Choceň
  - Litnea s.r.o. Neurologicka ambulance, Litoměřice
  - Neurosanatio s.r.o., Litomyšl
  - MP-neuro s.r.o. Poliklinika Modry pavilon, Ostrava
  - Nemocnice Pardubickeho kraje a.s. Pardubicka nemocnice Neurologická klinika, Pardubice
  - Diabetologicka ambulance Milan Kvapil s.r.o., Prague
  - Vestra Clinics s.r.o., Rychnov Nad Knežnou
- Hungary (6):
  - Budai Irgalmasrendi Korhaz Belgyógyászati Centrum, Budapest
  - Semmelweis Egyetem AOK I. sz. Belgyogyaszati Klinika, Budapest
  - Markhot Ferenc Oktatokorhaz es Rendelointezet Diabetesz Gondozo, Eger
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaz I. sz. Belgyogyaszati Osztaly, Gyula
  - Bacs-Kiskun Megyei Korhaz II. sz. Belgyogyaszati Osztaly, Kecskemét
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont I. Sz. Belgyogyaszati Klinika, Szeged
- Poland (7):
  - Silmedic Sp. z o.o., Katowice
  - Pro Familia Altera Sp. z o.o., Katowice
  - NZOZ Neuromed M. i M. Nastaj Sp. P., Lublin
  - RCMed Oddział Sochaczew, Sochaczew
  - Jeka Sławomir Niepubliczny Zakład Opieki Zdrowotnej "Nasz Lekarz" Praktyka Grupowa Lekarzy Rodzinnych z Przychodnia Specjalistyczna, Torun
  - NBR Polska Tomasz Klodawski, Warsaw
  - Medycyna Kliniczna, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lipone P, Ehler E, Nastaj M, Palka-Kisielowska I, Cruccu G, Truini A, Di Loreto G, Del Vecchio A, Pochiero I, Comandini A, Calisti F, Cattaneo A. Efficacy and Safety of Low Doses of Trazodone in Patients Affected by Painful Diabetic Neuropathy and Treated with Gabapentin: A Randomized Controlled Pilot Study. CNS Drugs. 2020 Nov;34(11):1177-1189. doi: 10.1007/s40263-020-00760-2. PMID 32936427
- See also: Sponsor's website — http://www.angelinipharma.com